CLINICAL TRIAL: NCT01259908
Title: Laparoscopic Aortic Surgery: Norwegian Experiance
Brief Title: Laparoscopic Surgical Treatment of Aorto-iliac Occlusive Disease
Acronym: LAS
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Sykehuset Ostfold (Other); Sorlandet Hospital HF (Other Government)
Responsible Party: Principal Investigator, Syed Sajid Hussain Kazmi, Consultant Surgeon, Oslo University Hospital
Other Study IDs: 2010/1953-4
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Aorto Iliac Occlusive Disease
Keywords: laparoscopic aortic surgery; aorto-iliac occlusive disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Laparoscopic vs open Ygraft: Patients with advanced atherosclerosis in aorto iliac segment operated with either laparoscopic aortobifemoral bypass or open aortobifemoral bypass shall be compared on the basis of the operative procedure for the primary endpoint, composite endpoint (all-cause mortality, systemic morbidity and graft thrombosis).
  Interventions: Procedure: Laparoscopic vs open Ygraft

INTERVENTIONS:
Procedure: Laparoscopic vs open Ygraft — Patients with aorto-iliac occlusive disease TASC type D operated with either laparoscopic aortobifemoral bypass or open aortobifemoral bypass shall be compared.

SUMMARY:
Patients with aorto-iliac occlusive disease (TASC, type D) operated with a totally laparoscopic aortobifemoral bypass operation and open aortobifemoral bypass operation will be followed up and the results will be compared between the two procedures on the basis of the primary endpoint, a composite endpoint defined as a combined incidence of systemic morbidity, graft thrombosis and all-cause mortality.

DETAILED DESCRIPTION:
Patients with aorto-iliac occlusive disease (TASC, type D) operated with a totally laparoscopic aortobifemoral bypass operation and open aortobifemoral bypass operation will be followed up and the results will be compared between the two procedures on the basis of the primary endpoint, a composite endpoint defined as a combined incidence of systemic morbidity, graft thrombosis and all-cause mortality.

Secondary endpoints like length of hospital stay, operation time, bleeding time shall also be considered.

Besides short form- 36 (SF-36) shall be used for the evaluation of patients health related quality of life, preoperatively,1,3,and 6 months and 1 year post-operatively.

Early, midterm and long time results shall be followed.

ELIGIBILITY:
All patients with a TASC D lesion in the aorto-iliac segment not amenable to or previously unsuccessfully treated by endovascular approach.

Exclusion Criteria:

* Unsuitable for surgery due to general health status

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with aorto-iliac occlusive disease (Type D lesion according to the Trans Atlantic Intersociety Consensus TASC II)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-09; Primary Completion 2023-05 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Composite endpoint (All-cause mortality, graft occlusion and systemic morbidity) | 2005-2015
  Composite endpoint defined as all-cause mortality, systemic morbidity and graft thrombosis.
  In this prospective comparative cohort study 50 consecutive patients with type D atherosclerotic lesions in the aortoiliac segment were treated with laparoscopic aortobifemoral bypass operation. The group was compared with 30 patients operated with open aortobifemoral bypass operations for the same disease and period of time. The groups were compared on the basis of composite endpoint All-cause mortality, graft occlusion and systemic morbidity). Stratification analysis was performed by using Mantel-Haenszel method with the patient time model. Cox multivariate regression method was used to adjust for confounding effect after considering the proportional hazard assumption. Cox proportional cause-specific hazard regression model was used for competing risk endpoints. Comparison of survival curves was done with the help of log- rank test.

SECONDARY OUTCOMES:
Operative time, operative bleeding, length of hospital stay, quality of life | 2005-2015
  Linear regression model was used to control for the confounding effect of the secondary continuous outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Background] Kazmi SS, Jorgensen JJ, Sundhagen JO, Krog AH, Florenes TL, Kolleros D, Abdelnoor M. A comparative cohort study of totally laparoscopic and open aortobifemoral bypass for the treatment of advanced atherosclerosis. Vasc Health Risk Manag. 2015 Sep 18;11:541-7. doi: 10.2147/VHRM.S92671. eCollection 2015. PMID 26425098
- [Background] Kazmi SS, Krog AH, Berge ST, Sundhagen JO, Sahba M, Falk RS. Patient-perceived health-related quality of life before and after laparoscopic aortobifemoral bypass. Vasc Health Risk Manag. 2017 May 12;13:169-176. doi: 10.2147/VHRM.S134669. eCollection 2017. PMID 28546754